CLINICAL TRIAL: NCT05171075
Title: A Multicenter, Randomized, Open-label, Blinded Endpoint Evaluation, Phase 3 Study Comparing the Effect of Abelacimab vs. Dalteparin on Venous Thromboembolism (VTE) Recurrence and Bleeding in Patients With GI/GU Associated VTE
Brief Title: A Study Comparing Abelacimab to Dalteparin in the Treatment of Gastrointestinal/Genitourinary Cancer and Associated VTE
Acronym: MAGNOLIA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Anthos Therapeutics, Inc. (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANT-008; 2021-003085-12 (EudraCT Number); CMAA868D12301 (Other: Novartis code)
Record Dates: First submitted 2021-11-22; First posted 2021-12-28 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Venous Thromboembolism; Deep Venous Thrombosis; Pulmonary Embolism
Keywords: Anticoagulants; VTE recurrence rate; PROBE design; LMWH; CAT; Cancer associated VTE; GI cancer; Abelacimab; Dalteparin; GU cancer; FXI; Major bleeding events; CRNM bleeding events
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism; Gastrointestinal Neoplasms | interventions — abelacimab; MAA868; Dalteparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abelacimab (Experimental): Abelacimab intravenous administration followed by monthly administration of the same dose subcutaneously
  Interventions: Biological: Abelacimab
- Dalteparin (Active Comparator): Dalteparin administered subcutaneously daily
  Interventions: Drug: Dalteparin

INTERVENTIONS:
Biological: Abelacimab — Abelacimab 150 mg
  Other Names: MAA868
  Arms: Abelacimab
Drug: Dalteparin — Dalteparin 200 IU/kg/day followed by 150 IU/kg/day
  Other Names: Fragmin
  Arms: Dalteparin

SUMMARY:
This is a Phase 3, multicenter, open-label, blinded endpoint study to evaluate the effect of abelacimab relative to dalteparin on venous thromboembolism (VTE) recurrence and bleeding in patients with gastrointestinal (GI)/genitourinary (GU) cancer associated VTE (Magnolia)

DETAILED DESCRIPTION:
Cancer associated thrombosis (CAT) is a severe medical condition which is characterized by high incidence of Venous thromboembolism (VTE) recurrence and high risk for bleeding. Patients with intact GI and GU cancer have increased bleeding risk with oral direct anticoagulants (DOACs), Guidelines advice caution with those DOACs or state preference for low molecular weight heparin (LMWH) in this population. The ANT-008 study will compare treatment with abelacimab monthly administration to LMWH daily subcutaneous (sc) administration over 6-month treatment. The study outcomes include VTE recurrence, bleeding event and treatment discontinuation at 6 months

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥18 years old or other legal maturity age according to the country of residence
* Confirmed GI (colorectal, pancreatic, gastric, esophageal, gastro-esophageal junction or hepatobiliary) or confirmed GU (renal, ureteral, bladder, prostate, or urethra) cancers if:

  * Unresectable, locally advanced, metastatic, or non-metastatic GI/GU cancer and
  * No intended curative surgery during the study
* Confirmed symptomatic or incidental proximal lower limb deep vein thrombosis (DVT) (i.e., popliteal, femoral, iliac, and/or inferior vena cava vein thrombosis) and/or a confirmed symptomatic pulmonary embolism (PE), or an incidental PE in a segmental, or larger pulmonary artery. Patients are eligible within 120 hours from diagnosis of the qualifying VTE.
* Anticoagulation therapy with LMWH for at least 6 months is indicated
* Able to provide written informed consent

Exclusion Criteria:

* Thrombectomy, insertion of a caval filter, or use of a fibrinolytic agent to treat the current (index) occurrence of DVT and/or PE
* More than 120 hours of pre-treatment with therapeutic doses of UFH, LMWH, or other anticoagulants
* An indication to continue treatment with therapeutic doses of an anticoagulant other than for VTE treatment prior to randomization (e.g., atrial fibrillation, mechanical heart valve, prior VTE)
* PE leading to hemodynamic instability (systolic BP <90 mmHg or shock).
* Acute ischemic or hemorrhagic stroke or intracranial hemorrhage, in the last 4 weeks preceding screening.
* Brain trauma, or cerebral or a spinal cord surgery or spinal procedures such as lumbar puncture or epidural/spinal anesthesia within 4 weeks of screening
* Need for aspirin in a dosage of more than 100 mg/day or, any other antiplatelet agent alone or in combination with aspirin
* Bleeding requiring medical attention at the time of randomization or in the preceding 4 weeks
* Planned brain, spinal cord, cardiac, vascular, major thoracic and/or major abdominal surgery in the 4 weeks following randomization
* History of heparin induced thrombocytopenia
* Infective acute or subacute endocarditis at the time of presentation
* Primary brain cancer or untreated intracranial metastasis
* Eastern Cooperative Oncology Group (ECOG) performance status of 3 or 4 at screening
* Life expectancy of <3 months at randomization
* Calculated creatinine clearance (CrCl) <30 mL/min at the screening visit
* Platelet count <50,000/ mm3 at the screening visit
* Hemoglobin <8 g/dL at the screening visit
* Acute hepatitis, chronic active hepatitis, liver cirrhosis; or an alanine aminotransferase ≥3 times and/or bilirubin ≥2 times the upper limit of normal (ULN) at the screening visit in the absence of clinical explanation
* Uncontrolled hypertension (systolic blood pressure [BP] > 180 mm Hg or diastolic BP >100 mm Hg despite antihypertensive treatment)
* Women of child-bearing potential (WOCBP) who are unwilling or unable to use highly effective contraceptive measures during the study from screening up to 3 days after last treatment of dalteparin or 100 days after administration of abelacimab
* Sexually active males with sexual partners of childbearing potential must agree to use a condom or other reliable contraceptive measure up to 3 days after last treatment of dalteparin or 100 days after administration of abelacimab
* Pregnant or breast-feeding women
* History of hypersensitivity to any of the study drugs (including dalteparin) or its excipients, to drugs of similar chemical classes, or any contraindication listed in the label for dalteparin
* Subjects with any condition that in the judgement of the Investigator would place the subject at increased risk of harm if he/she participated in the study
* Use of other investigational (not-registered) drugs within 5 half-lives prior to enrollment or until the expected pharmacodynamic effect has returned to baseline, whichever is longer. Participation in academic non-interventional studies or interventional studies, comprising testing different strategies or different combinations of registered drugs is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Time to first event of centrally adjudicated VTE recurrence | up to 6 months
  Time to first adjudicated venous thromboembolism (VTE) event recurrence

SECONDARY OUTCOMES:
Time to first event of ISTH-adjudicated major or clinically relevant non-major (CRNM) bleeding events | up to 6 months
  Time to first adjudicated major or clinically relevant non-major (CRNM) bleeding event
Time to first event of VTE recurrence, ISTH adjudicated major or ISTH-adjudicated CRNM bleeding events | up to 6 months
  Time to first adjudicated venous thromboembolism (VTE) or bleeding event
Time to event of permanent treatment discontinuation not due to death | up to 6 months
  Time to permanent discontinuation not due to death
Time to first event of ISTH-adjudicated CRNM bleeding events | up to 6 months
  Time to first adjudicated clinically relevant non-major (CRNM) bleeding event
Time to first event of ISTH-adjudicated major bleeding events | Up to 6 months
  Time to first adjudicated major bleeding event
Time to first event of GI ISTH-adjudicated major and GI CRNM bleeding events | up to 6 months
  Time to first adjudicated gastrointestinal (GI) major and clinically relevant non-major (CRNM) bleeding event
All-cause death, vascular death, serious adverse events, adverse events leading to drug discontinuation, other adverse events, abnormal lab tests, etc. presented as rate per 100 patient-years | up to 6 months
For patients treated with abelacimab: percent with injection site reactions/severity, hypersensitivity reactions/severity, anti-drug antibody formation, neutralizing antibody | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (116):
- United States (10):
  - Washington DC VAMC, Washington D.C., District of Columbia
  - NorthShore University Health System, Evanston, Illinois
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center-Middletown, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center-Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center-West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
- Australia (3):
  - Blacktown Hospital, Blacktown, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Northern Health, Epping, Victoria
- Austria (2):
  - LK Wiener Neustadt, Neustadt
  - Medical University of Vienna, Vienna
- Canada (5):
  - Hamilton Health Sciences, Juravinski Hospital and Cancer Centre, Hamilton, Ontario
  - Ottawa Hospital Research Instituite, Ottawa, Ontario
  - University of Calgary, Calgary
  - Sault Area Hospital, Marie
  - Toronto General Hospital, Toronto
- China (13):
  - Beijing Shijitan Hosp., Beijing
  - Peking University Third Hospital, Beijing
  - Jilin Province Tumor Hospital, Ch’ang-ch’un
  - Southern Medical University - Zhujiang Hospital, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - The Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou
  - Huizhou Municipal Central Hospital, Huizhou
  - Nanjing First Hospital, Nanjing
  - Nantong Tumor Hospital (Tumor Hospital Affiliated to Nantong University ), Tongzhou
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Union Hospital Tongji Medical College Huazhong University of Science &Technology, Wuhan
  - Hubei Cancer Hospital, Wuhan
  - The Second Hospital of Jiaxing, Zhejiang
- Czechia (4):
  - Masarykuv onkologicky ustav, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - Onkologická klinika VFN a 1. LF UK, Prague
  - Thomayerova nemocnice, Prague
- France (16):
  - CHU de Limoges - Hôpital Dupuytren, Limoges, Cedex
  - CH Le Puy en Velay, Le Puy-en-Velay, Chantemesse
  - Hôpital Louis Mourier, Colombes, Renouiflers
  - CHU de Nancy - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy, Rue Du Morvan
  - Nouvel Hôpital Civil de Strasbourg, Strasbourg, Strasbourg
  - CHU Angers - Hôpital Hôtel Dieu, Angers
  - CHU Clermont Ferrand - Hopital Gabriel Montpied, Clermont-Ferrand
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hospices Civils de Lyon (HCL) - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - CHU de Rouen - Hôpital de Bois Guillaume, Rouen
  - CHU de Saint-Etienne - Hopital Nord, Saint-Etienne
  - CHU Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - Centre Hospitalier Intercommunal de Toulon, Toulon
  - CHU de Nancy - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy
- Germany (5):
  - Staedtisches Klinikum Dresden Standort Dresden-Friedrichstadt, Dresden
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Praxis für Gefäßmedizin, Görlitz
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinik Leipzig, Leipzig
- Hungary (2):
  - Debreceni Egyetem, Debrecen
  - Markhot Ferenc Oktatokorhaz es Rendelointezet, Eger
- Ireland (3):
  - Cork University Hospital, Cork
  - Bon Secour Hospital, Cork
  - Beaumont Hospital, Dublin
- Italy (13):
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - Arcispedale S. Maria Nuova Azienda Ospedaliera di Reggio Emilia, Bologna
  - Presidio Ospedaliero di Castelfranco Veneto, Castelfranco Veneto
  - SS. ma Annunziata, Chieti
  - Ospedale Civile Dell Annunziata, Cosenza
  - Ospedale Degli Infermi, Faenza
  - Azienda Socio Sanitaria Territoriale Santi Paolo e Carlo, Milan
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - Azienda Ospedale - Università Padova, Padua
  - Ospedale Universitario, Padua
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Ospedale San Bortolo di Vicenza, Vicenza
- Latvia (3):
  - Daugavpils Regional Hospital, Daugavpils
  - Liepaja Regional Hospital, Liepāja
  - Pauls Stradins CUH, Riga
- Netherlands (8):
  - Meander Medisch Centrum, Amersfoort
  - Albert Schweitzer Ziekenhuis, Dordwijk, Dordrecht
  - Spaarne Gasthuis (Kennemer Gasthuis) - Haarlem-Zuid, Haarlem
  - Amsterdam University Medical Center, Holland
  - Leids Universitair Medisch Centrum, Leiden
  - Radboud Universitair Medisch Centrum, Nijmegen
  - Ikazia Ziekenhuis, Rotterdam
  - Haga Ziekenhuis, The Hague
- Norway (2):
  - Østfold Hospital Kalnes, Fredrikstad
  - Akershus Univeristy Hospital, Lørenskog
- South Korea (3):
  - Jeonbuk National University Hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam
  - Ewha Womans University Mokdong Hospital, Seoul
- Spain (16):
  - Hospital Universitario Del Vinalopo, Alicante
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Ciudad de Jaen, Jaén
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Clinica Universidad de Navarra, Madrid
  - MD Anderson Cancer Centre, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Complejo Hospitalario Universitario de Ourense, Ourense
  - Hospital Universitario Central de Asturia, Oviedo
  - Clinica Universidad de Navarra, Pamplona
  - Corporacio Sanitaria Parc Tauli, Sabadell
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville
- Länssjukhuset Sundsvall-Härnösand, Sundsvall, Sweden
- Hopital Universitaire Geneve, Geneva, Switzerland
- Taiwan (3):
  - Far Eastern Memorial Hospital, New Taipei City
  - National Cheng Kung University (NCKU) Hospital, Tainan
  - Tri-Service General Hospital, Taipei
- United Kingdom (3):
  - University Hospital of Wales, Cardiff, England
  - Castle Hill Hospital, Department of Oncology & Haematology, Cottingham, ENG
  - The Newcastle Upon Tyne Hospitals, Newcastle upon Tyne, ENG

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com